CLINICAL TRIAL: NCT03258463
Title: Travelling for Rights
Acronym: TOR
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 16-006
Record Dates: First submitted 2017-08-17; First posted 2017-08-23 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy Termination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Time Period 1: Women who obtained an abortion from January 1 2012-December 31 2012
- Time Period 2: Women who obtained an abortion from May 1 2014-April 30 2015.
  Interventions: Other: Change in Texas Law

INTERVENTIONS:
Other: Change in Texas Law — The change in Texan laws occurring from July 2013-January 2014
  Groups: Time Period 2

SUMMARY:
This will be a retrospective cohort study comparing women obtaining an abortion in New Mexico and living in Texas and women obtaining an abortion in New Mexico and living in New Mexico .

DETAILED DESCRIPTION:
This will be a retrospective cohort study comparing women obtaining an abortion in New Mexico and living in Texas and women obtaining an abortion in New Mexico and living in New Mexico in two different time periods (time period #1 is from January 1 2012-December 31 2012 and time period #2 is from May 1 2014-April 30 2015. Our exposure is a state in which a woman lives in (New Mexico or Texas). Our intervention is the change in Texan laws occurring from July 2013-January 2014.

ELIGIBILITY:
Inclusion Criteria:

* Women obtaining an induced abortion at one of the following clinics:

University of New Mexico's Center for Reproductive Health (UNM CRH), Planned Parenthood - Albuquerque Surgical Center or Southwestern Women's Options.

* Women residing in Texas or New Mexico. -Women obtaining an induced abortion between January 1 2012-

Exclusion Criteria:

* No chart available for data extraction
* Gestational age at time of abortion initiation ≥ 24 weeks gestation as determined by ultrasound imaging.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Charts of women obtaining an induced abortion.
Sampling Method: Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Proportion of women from Texas travelling to NM, to obtain an abortion. | 2012-2015
  The primary objective of this study is to determine whether the proportion of Texan women obtaining an induced abortion in New Mexico increased between time period #1 and time period #2.

CONTACTS AND LOCATIONS:
Overall Officials: Eve Epsey, MD, MPH, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States